CLINICAL TRIAL: NCT04302701
Title: Patching Versus Dichoptic Stimulation Using Virtual Reality in Anisometropic Amblyopia
Brief Title: Dichoptic Treatment vs. Patching for Moderate Anisometropic Amblyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Professor of Ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dichoptic-123
Record Dates: First submitted 2020-01-02; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Amblyopia; Anisometropia
MeSH Terms: conditions — Amblyopia; Anisometropia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dichoptic arm (Experimental): Dichoptic visual training will be performed with the patient wearing his spectacles using the computer game included in Vivid Vision (Vivid Vision, San Francisco, USA) which will be run in the Oculus Rift OC CV1 virtual reality head mounted display (Oculus VR, Menlo Park, California, USA). Each subject will have 20 treatment sessions, divided into 1 hour-sessions performed twice a week for 10 weeks. Each session will be 60 minutes. Adherence to the treatment regimen will be assessed by the number of hours spent in training at the end of 5th week.
  Interventions: Other: Dichoptic treatment using virtual reality
- Patching (Active Comparator): Patients in the control group will be instructed to continue wearing spectacles if required. Patients will be prescribed two continuous hours of daily patching with at least one hour of near activities during patching. Adhesive skin patches will be provided by the study. The parent/patient will be instructed to spend at least one of the hours of patching time each day performing eye-hand coordination activities at near. Adherence to the treatment protocol will be assessed by having the parent call / send a message to an investigator at the start and end of the occlusion sessions completed each day, thus making the most as accurate as possible assessment of the patient's adherence to the prescribed treatment
  Interventions: Other: Patching

INTERVENTIONS:
Other: Dichoptic treatment using virtual reality — Dichoptic visual training will be performed with the patient wearing his spectacles using the computer game included in Vivid Vision (Vivid Vision, San Francisco, USA) which will be run in the Oculus Rift OC CV1 virtual reality head mounted display (Oculus VR, Menlo Park, California, USA). Each subject will have 20 treatment sessions, divided into 1 hour-sessions performed twice a week for 10 weeks. Each session will be 60 minutes. Adherence to the treatment regimen will be assessed by the number of hours spent in training at the end of 5th week.
  Arms: Dichoptic arm
Other: Patching — Patients in the control group will be instructed to continue wearing spectacles if required. Patients will be prescribed two continuous hours of daily patching with at least one hour of near activities during patching. Adhesive skin patches will be provided by the study. The parent/patient will be instructed to spend at least one of the hours of patching time each day performing eye-hand coordination activities at near.
  Arms: Patching

SUMMARY:
Recently, there has been an increased interest in evaluating binocular therapies (e.g perceptual learning and dichoptic treatment) for amblyopia. They are designed to improve amblyopia through binocular stimulation by unlocking binocular visual function. The objective of the study is to compare the visual and sensory outcome of 2-hour patching to dichoptic stimulation using virtual reality head mounted display in the management of patients with moderate anisometropic amblyopia. The investigators will include children older than 6 years and adults up to the age of thirty five years with anisometropic amblyopia who either had no prior treatment for amblyopia or had prior treatment for amblyopia using patching therapy but with residual amblyopia defined as >= 0.3 logMAR lines between the best-corrected visual acuity in the sound eye and in the amblyopic eye and with moderate amblyopia in the more anisometropic eye defined as best-corrected visual acuity better than 6/60 but =< 6/18. Patients will be randomized into 2 groups according to age using stratified randomization:

* Group P: (Patching Group): This group will have 2 hours of patching each day for 10 weeks.
* Group D (Dichoptic Group): This group will have 1 hour of dichoptic stimulation using the virtual reality system twice a week for 10 weeks for a total of 20 hours of training.

DETAILED DESCRIPTION:
The investigators are planning to conduct a study to compare the visual and sensory outcome of 2-hour patching to dichoptic stimulation using virtual reality head mounted display in the management of patients with moderate anisometropic amblyopia. This is a randomized clinical trial. The investigators will include children older than 6 years and adults up to the age of thirty five years with anisometropic amblyopia who either had no prior treatment for amblyopia or had prior treatment for amblyopia using patching therapy but with residual amblyopia defined as >= 0.3 logMAR lines between the best-corrected visual acuity in the sound eye and in the amblyopic eye and with moderate amblyopia in the more anisometropic eye defined as best-corrected visual acuity better than 6/60 but =< 6/18.n Recruitment will occur from the Ophthalmology Outpatient Clinics in Kasr El-Ainy Hospital.

Eligible patients who agree to participate in the study will undergo a 1-hour trial session of dichoptic stimulation using the same head-mounted virtual reality system that will be used in the study to ensure that the patient can use the system. Only patients who are able to understand and to complete the 1-hour session will be enrolled in the study.

Patients will be randomized into 2 groups according to age using stratified randomization:

* Group P: (Patching Group): This group will have 2 hours of patching each day for 10 weeks.
* Group D (Dichoptic Group): This group will have 1 hour of dichoptic stimulation using the virtual reality system twice a week for 10 weeks for a total of 20 hours of training.

Patients will be further subdivided into 2 subgroups according to whether prior patching therapy has been done and failed, or the patient has never received any form of patching therapy. The difference in the outcomes in both subgroups will be analyzed separately.

All patients will have a baseline ophthalmological examination including visual acuity testing, manifest and cycloplegic refraction, slit lamp examination with funduscopy, cover test and worth four dot test. Best corrected visual acuity (BCVA) will be measured using a single crowded letter in an ETDRS chart mounted on a computer display projector. The stereoacuity will be measured using the TNO test. The motor alignment will be evaluated using prism and alternating cover test at 6 meters and at 33 cm. BCVA and stereoacuity will be measured before and after 10 weeks of treatment. Then, they will be re-measured 10 weeks after the cessation of both treatments to assess their long-term effects. All measurements will be taken by an investigator who will be masked to the study design.

Dichoptic treatment group: Dichoptic visual training will be performed with the patient wearing his spectacles using the computer game included in Vivid Vision (Vivid Vision, San Francisco, USA) which will be run in the Oculus Rift OC CV1 virtual reality head mounted display (Oculus VR, Menlo Park, California, USA). Each subject will have 20 treatment sessions, divided into 1 hour-sessions performed twice a week for 10 weeks. Each session will be 60 minutes. Adherence to the treatment regimen will be assessed by the number of hours spent in training at the end of 5th week.

Patching group: Patients in the control group will be instructed to continue wearing spectacles if required. Patients will be prescribed two continuous hours of daily patching with at least one hour of near activities during patching. Adhesive skin patches will be provided by the study. The parent/patient will be instructed to spend at least one of the hours of patching time each day performing eye-hand coordination activities at near. Adherence to the treatment protocol will be assessed by having the parent call / send a message to an investigator at the start and end of the occlusion sessions completed each day, thus making the most as accurate as possible assessment of the patient's adherence to the prescribed treatment. Written consent will be obtained by either the principal investigator or other investigators in the study. Adverse events will include any sense of dizziness, vertigo, or diplopia at any time and will be tabulated and reported at the end of each week. The data will be collected with privacy and confidentiality as patients will be allocated ID numbers and data will be analyzed accordingly.

A sample size of 38 participants in each group will be selected to have 90% power with a 2-sided type I error of 5% to detect a treatment group difference at 10 weeks if the true difference in the mean gain of new letters was 3.75, assuming a standard deviation (SD) of change of 5 letters, based on a prior PEDIG study. Assuming a 10% drop-out rate, a total of 42 patients in each group will need to be recruited.

Comparison between both groups will be done using independent t-test for continuous variables and Fisher Exact test for categorical variables. Analyses for secondary outcomes of visual acuity and stereoacuity will be adjusted for multiple testing using the Bonferroni method such that the overall type I error rate will be 5% within the 2sets of secondary outcomes. Exploratory analyses will be conducted for secondary outcomes and adherence measures for participants assigned to control treatment who later received 10 weeks of binocular treatment. Log file data at 5 weeks and 10 weeks will be used to quantify measures of adherence (treatment duration and change in contrast presented to the fellow eye) and to examine the relationship between these adherence measures and treatment response. For each participant, the total hours of completed and prescribed game play will be calculated, and the percentage of prescribed treatment completed (adherence) will be computed using the ratio of the completed and prescribed hours of game play for that interval. Analyses will be conducted using SAS version 9.4 (SAS Inc, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with anisometropic amblyopia who had proper optical correction using spectacles or contact lenses for the past 6 weeks. Anisometropic amblyopia will be defined as difference > 0.3 logMAR lines in best-corrected visual acuity with difference in the spherical equivalent of both eyes > 1 D, in the absence of other causes for amblyopia such as organic causes, or manifest strabismus < 5 PD by simultaneous prism and cover test. Patients will be included in the study only if they had no treatment for amblyopia for the past month other than spectacles and/or contact lenses.

Exclusion Criteria:

* Patients with development delay
* Prior ocular surgery
* Co-existing ocular disease
* Patients with allergy to patch material
* History of problems with prior use of virtual reality systems

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity at 10 weeks | 10 weeks
  Change in amblyopic eye VA letter score from baseline to 10 weeks.

SECONDARY OUTCOMES:
Compliance to treatment | 10 weeks
  Average number of hours of completed treatment in both groups defined as number of hours of completed dichoptic treatment in the dichootic group and number of hours of patching as self reported by patients in the patching group
Number of patients developing misalignment | 10 weeks
  Number of patients developing misalignment after 10 weeks of therapy will be assessed
Regression of amblyopic eye visual acuity | 20 weeks
  Amblyopic eye visual acuity letter score 10 weeks after cessation of treatments
Changes in visual acuity in the sound eye | 10 weeks
  Change in sound eye VA letter score from baseline to 10 weeks.
Changes in near stereopsis | 10 weeks
  Stereopsis using TNO test will be assessed

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after 3 years
Access Criteria: The principal investigator will review requests for information.

REFERENCES:
- [Background] Holmes JM, Kraker RT, Beck RW, Birch EE, Cotter SA, Everett DF, Hertle RW, Quinn GE, Repka MX, Scheiman MM, Wallace DK; Pediatric Eye Disease Investigator Group. A randomized trial of prescribed patching regimens for treatment of severe amblyopia in children. Ophthalmology. 2003 Nov;110(11):2075-87. doi: 10.1016/j.ophtha.2003.08.001. PMID 14597512
- [Background] Hess RF, Thompson B, Baker DH. Binocular vision in amblyopia: structure, suppression and plasticity. Ophthalmic Physiol Opt. 2014 Mar;34(2):146-62. doi: 10.1111/opo.12123. PMID 24588532
- [Background] Polat U, Ma-Naim T, Spierer A. Treatment of children with amblyopia by perceptual learning. Vision Res. 2009 Oct;49(21):2599-603. doi: 10.1016/j.visres.2009.07.008. Epub 2009 Jul 19. PMID 19622368
- [Background] Manh VM, Holmes JM, Lazar EL, Kraker RT, Wallace DK, Kulp MT, Galvin JA, Shah BK, Davis PL; Pediatric Eye Disease Investigator Group. A Randomized Trial of a Binocular iPad Game Versus Part-Time Patching in Children Aged 13 to 16 Years With Amblyopia. Am J Ophthalmol. 2018 Feb;186:104-115. doi: 10.1016/j.ajo.2017.11.017. Epub 2017 Nov 28. PMID 29196184
- [Background] Li SL, Reynaud A, Hess RF, Wang YZ, Jost RM, Morale SE, De La Cruz A, Dao L, Stager D Jr, Birch EE. Dichoptic movie viewing treats childhood amblyopia. J AAPOS. 2015 Oct;19(5):401-5. doi: 10.1016/j.jaapos.2015.08.003. PMID 26486019
- [Background] Ziak P, Holm A, Halicka J, Mojzis P, Pinero DP. Amblyopia treatment of adults with dichoptic training using the virtual reality oculus rift head mounted display: preliminary results. BMC Ophthalmol. 2017 Jun 28;17(1):105. doi: 10.1186/s12886-017-0501-8. PMID 28659140
- See also: The link to the software of the VR games used in this study — https://www.seevividly.com/